CLINICAL TRIAL: NCT01439854
Title: Regulation of Hepatic and Peripheral Glucose Metabolism: Protocol IVA. Effect of Plasma Glucose Reduction by Selective SLGT2 Inhibition on Mitochondrial Dysfunction and Impaired Insulin Signaling/Sensitivity in T2DM
Brief Title: Study of Dapagliflozin on Mitochondrial Dysfunction and Impaired Insulin Signaling/Action
Acronym: DAPA MITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5 R01 DK024092-27/NIH Prot IV; R01DK024092 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-09-23 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Insulin Sensitivity; Multiple Mitochondrial Dysfunctions Syndrome
Keywords: Insulin sensitivity; Mitochondrial function; Glucose toxicity; Glucosuria
MeSH Terms: conditions — Insulin Resistance; Multiple Mitochondrial Dysfunctions Syndrome; Glycosuria | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): this arm is control
  Interventions: Drug: Placebo
- Dapagliflozin (Experimental): Interventional arm
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Treatment arm, 10 mg per day for 2 weeks
  Arms: Dapagliflozin
Drug: Placebo — Patients are treated with placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of the chronic treatment of type 2 diabetes (T2DM) with dapagliflozin on: (1) mitochondrial gene function/expression and insulin signaling/action and (2) oral glucose tolerance and beta cell function. Dapagliflozin is a potent, highly specific inhibitor of renal glucose transport [SGLT2].

DETAILED DESCRIPTION:
"Glucotoxicity" has been implicated as a cause of insulin resistance and impaired beta cell function in T2DM. Abundant support for the glucotoxicity hypothesis has been provided by in vivo and in vitro studies in animals, but a rigorous test of this hypothesis in man is lacking. The investigators propose to test the glucotoxicity hypothesis by chronically reducing the plasma glucose in type 2 diabetic subjects (T2DM) with an inhibitor of renal glucose transport, dapaglifozin, and examining the effect of restoration of normoglycemia on mitochondrial function and insulin signaling/sensitivity. Lastly, the investigators will test the "glucolipotoxicity" hypothesis, which states that the toxic effects of elevated plasma FFA on insulin sensitive tissues (i.e., muscle) are magnified in the presence of concurrent hyperglycemia. Thus, high glucose levels increase malonyl CoA, which inhibits CPT I, leading to accumulation of FACoA/DAG, which impair mitochondrial function and inhibit insulin action.

ELIGIBILITY:
Inclusion Criteria:

* T2DM
* Drug Naive Or On Oral Therapy

Exclusion Criteria:

* Insulin Treatment
* Major Organ Disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Devjit Tripathy, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Diabetes Division, UTHSCSA, San Antonio, Texas, United States

REFERENCES:
- [Result] Daniele G, Xiong J, Solis-Herrera C, Merovci A, Eldor R, Tripathy D, DeFronzo RA, Norton L, Abdul-Ghani M. Dapagliflozin Enhances Fat Oxidation and Ketone Production in Patients With Type 2 Diabetes. Diabetes Care. 2016 Nov;39(11):2036-2041. doi: 10.2337/dc15-2688. Epub 2016 Aug 25. PMID 27561923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (2.1) | 51.9 (2.3) | 53.6 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (1.5) | 30.9 (1.8) | 31.8 (1.7)
A1C (average blood glucose level over 3 months [Mean (Standard Deviation); unit: percentage] | 8.7 (0.4) | 8.5 (0.4) | 8.6 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity
Description: The change in insulin sensitivity and total glucose disposal measured at two weeks with the insulin clamp compared to baseline. This is measured using TGD (whole body tissue glucose disposal)/SSPI (steady state plasma insulin concentration) ratio
Time Frame: baseline, two weeks
Measure: Mean (Standard Deviation); unit: mg/kg.min per µU/ml
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 8 | 10
mg/kg.min per µU/ml
  Baseline Measurement | 3.18 (0.51) | 3.85 (0.71)
  2 weeks | 3.57 (0.51) | 5.22 (0.56)

2. Secondary Outcome: Change in Mitochondrial Function
Description: The change in mitochondrial function/gene expression at two weeks compared to baseline. This was measured by energy expenditure.
Time Frame: baseline, two weeks
Measure: Mean (Standard Deviation); unit: cal/min.kg
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 8 | 10
cal/min.kg
  Baseline Measurement | 1.06 (0.1) | 1.3 (0.1)
  Measurement at 2 weeks | 1.0 (0.1) | 1.34 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse events are collected over a 2 week period
Arm/Group | Placebo | Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT01439854/Prot_SAP_000.pdf